CLINICAL TRIAL: NCT04438031
Title: Evaluation of the Navigation Prevention Program: Durham
Brief Title: Navigation Study: Durham
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104042
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Prenatal; Postnatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Navigation Intervention Prenatal 1.0 (arm closed and modified to 2.0 design. Data will not be used) (Experimental): This program recruits mothers in OB/GYN (prenatal) offices, provides up to three Navigation visits (using prenatal navigation version 1.0), establishes connections between the family and primary health care or other community providers, and then follows up one month later to confirm these referrals. Navigators will assess and support family needs across multiple developmentally-appropriate domains at each age. Prenatally, the domains include support for (1) health and access to healthcare, (2) adjustments to pregnancy, (3) household and material needs, and (4) family safety. At 12, 24, and 36 months, the domains include support for (1) child basic needs, (2) parenting and child behavior, (3) child health and development, and (4) parent health and well-being.
  Interventions: Behavioral: Navigation Intervention Prenatal 1.0 (intervention discontinued, modified to 2.0. Data will not be used)
- Control Intervention (Other): Brief educational information will be provided about pregnancy (provided prenatally) and child development at 12, 24, and 36 months.
  Interventions: Behavioral: Control Intervention
- Navigation Intervention Prenatal 2.0 (Experimental): This program recruits mothers in OB/GYN offices. Mothers are offered visits from a Navigator prenatally and postnatally (12-, 24-, and 36-months). During visits, the Navigator works with the mother to identify family needs, establishes connections between the family and community providers, and follows up one month later to confirm these referrals. Navigators assess and support family needs across 13 factors: caregiver health, infant health, healthcare plans, childcare plans, parent-child relationship, management of infant crying/behavior, household safety/material supports, family/community violence, history of parenting difficulties, parent well-being, substance use, parent emotional support, and other needs not related to first 12 factors. Navigation 2.0 is a revision of 1.0 in which adjustments to the protocol were made to improve guidance for Community Navigators and aid their assessments of family needs.
  Interventions: Behavioral: Navigation Intervention Prenatal 2.0

INTERVENTIONS:
Behavioral: Navigation Intervention Prenatal 1.0 (intervention discontinued, modified to 2.0. Data will not be used) — This program recruits mothers in OB/GYN (prenatal) offices, provides up to three Navigation visits (using prenatal navigation version 1.0), establishes connections between the family and primary health care or other community providers, and then follows up one month later to confirm these referrals. Navigators will assess and support family needs across multiple developmentally-appropriate domains at each age. Prenatally, the domains include support for (1) health and access to healthcare, (2) adjustments to pregnancy, (3) household and material needs, and (4) family safety. At 12, 24, and 36 months, the domains include support for (1) child basic needs, (2) parenting and child behavior, (3) child health and development, and (4) parent health and well-being.
  Arms: Navigation Intervention Prenatal 1.0 (arm closed and modified to 2.0 design. Data will not be used)
Behavioral: Control Intervention — Brief information will be provided about pregnancy prenatally and child development at 12, 24, and 36 months.
  Arms: Control Intervention
Behavioral: Navigation Intervention Prenatal 2.0 — This program recruits mothers in OB/GYN offices. Mothers are offered visits from a Navigator prenatally and postnatally (12-, 24-, and 36-months). During visits, the Navigator works with the mother to identify family needs, establishes connections between the family and community providers, and follows up one month later to confirm these referrals. Navigators assess and support family needs across 13 factors: caregiver health, infant health, healthcare plans, childcare plans, parent-child relationship, management of infant crying/behavior, household safety/material supports, family/community violence, history of parenting difficulties, parent well-being, substance use, parent emotional support, and other needs not related to first 12 factors. Navigation 2.0 is a revision of 1.0 in which adjustments to the protocol were made to improve guidance for Community Navigators and aid their assessments of family needs.
  Arms: Navigation Intervention Prenatal 2.0

SUMMARY:
The purpose of the proposed study is to evaluate the implementation and impact of a new, community-wide prevention program, "Navigation", on maternal and infant health and well-being. This program recruits mothers at the OB/GYN or pediatrician's office and provides up to several visits (prenatally, 12 months, 24 months, and 36 months) to assess family needs, establishes connections between the family and primary health care or other community providers, and then follows up one month later to confirm these referrals.

DETAILED DESCRIPTION:
Of note, 400 families were enrolled under Navigation 1.0, however, their data will not be included in any analysis due to the design changes (Navigation 2.0). The anticipated total of 800 subjects is specific to the 2.0 enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Families will be eligible for the study if they go to the certain OB/GYN offices (to be updated later) for their first prenatal visit
* Families will be eligible for the study if they go to the Roxboro Road Pediatric Care Practice for their child's 12-, 24-, or 36-month well visit
* Primary language is English or Spanish

Exclusion Criteria:

* Families residing outside of Durham County
* Families that are planning to move out of either county within the next 2 months at the time of recruitment
* Families will also be ineligible if the parent has a cognitive impairment that impairs their ability to consent/participate.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the implementation by the rate of enrollment in the Navigation program. | Prenatally (up until delivery of target child)
  Proportion of participants in the Navigation group who agree to schedule a prenatal Navigation visit, which will be collected from enrollment logs.
Evaluate the implementation by the rate of retention in the Navigation program. | 12 months
  This will be collected from participant tracking logs completed by the navigators (i.e., whether they completed the 12-month Navigation visit with the participant).
Evaluate the implementation by the rate of retention in the Navigation program. | 24 months
  This will be collected from participant tracking logs completed by the navigators (i.e., whether they completed the 24-month Navigation visit with the participant).
Evaluate the implementation by the rate of retention in the Navigation program. | 36 months
  This will be collected from participant tracking logs completed by the navigators (i.e., whether they completed the 36-month Navigation visit with the participant).
Evaluate the implementation by the fidelity of implementation of the Navigation manual by Navigators. | 12 months
  For 10% of the Navigation visits, a second Navigator will observe the primary Navigator. The second Navigator will check using a list of program elements from the program manual to assess whether the primary Navigator adheres to each program element. In addition, the second Navigator will score the family on each of the Navigation domains. Fidelity of implementation will be measure by the percent adherence to the program manual and the inter-rater reliability on the domain scores using Cohen's kappa statistic.
Evaluate the implementation by the fidelity of implementation of the Navigation manual by Navigators. | 24 months
  For 10% of the Navigation visits, a second Navigator will observe the primary Navigator. The second Navigator will check using a list of program elements from the program manual to assess whether the primary Navigator adheres to each program element. In addition, the second Navigator will score the family on each of the Navigation domains. Fidelity of implementation will be measure by the percent adherence to the program manual and the inter-rater reliability on the domain scores using Cohen's kappa statistic.
Evaluate the implementation by the fidelity of implementation of the Navigation manual by Navigators. | 36 months
  For 10% of the Navigation visits, a second Navigator will observe the primary Navigator. The second Navigator will check using a list of program elements from the program manual to assess whether the primary Navigator adheres to each program element. In addition, the second Navigator will score the family on each of the Navigation domains. Fidelity of implementation will be measure by the percent adherence to the program manual and the inter-rater reliability on the domain scores using Cohen's kappa statistic.
Evaluate the implementation by the proportion of families receiving screening scores that indicate risk for negative child and/or family outcomes. | Prenatal (before delivery of target child)
  This will be collected from case report forms completed by the Navigators. For each intervention domain of interest, Navigators will rate family needs on a 1-4 scale with scores of 3 and 4 indicating a need for referral to community resources. This outcome will be measured as the proportion of families receiving at least one score of 3 or 4.
Evaluate the implementation by the proportion of families receiving screening scores that indicate risk for negative child and/or family outcomes. | 12 months
  This will be collected from case report forms completed by the Navigators. For each intervention domain of interest, Navigators will rate family needs on a 1-4 scale with scores of 3 and 4 indicating a need for referral to community resources. This outcome will be measured as the proportion of families receiving at least one score of 3 or 4.
Evaluate the implementation by the proportion of families receiving screening scores that indicate risk for negative child and/or family outcomes. | 24 months
  This will be collected from case report forms completed by the Navigators. For each intervention domain of interest, Navigators will rate family needs on a 1-4 scale with scores of 3 and 4 indicating a need for referral to community resources. This outcome will be measured as the proportion of families receiving at least one score of 3 or 4.
Evaluate the implementation by the proportion of families receiving screening scores that indicate risk for negative child and/or family outcomes. | 36 months
  This will be collected from case report forms completed by the Navigators. For each intervention domain of interest, Navigators will rate family needs on a 1-4 scale with scores of 3 and 4 indicating a need for referral to community resources. This outcome will be measured as the proportion of families receiving at least one score of 3 or 4.
Evaluate the implementation by the proportion of families referred to community resources. | Prenatally (before delivery of target child)
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate any community resources to which they refer families. This outcome will be measured as the proportion of families that are referred to one or more community resources by the Navigator.
Evaluate the implementation by the proportion of families referred to community resources. | 12 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate any community resources to which they refer families. This outcome will be measured as the proportion of families that are referred to one or more community resources by the Navigator.
Evaluate the implementation by the proportion of families referred to community resources. | 24 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate any community resources to which they refer families. This outcome will be measured as the proportion of families that are referred to one or more community resources by the Navigator.
Evaluate the implementation by the proportion of families referred to community resources. | 36 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate any community resources to which they refer families. This outcome will be measured as the proportion of families that are referred to one or more community resources by the Navigator.
Evaluate the implementation by the proportion of families that initiate community services. | Prenatally (before delivery of target child)
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate whether families initiated participation in the community services to which they were referred, if any. This outcome will be measured as the proportion of families referred to community services that initiate participation in at lease one community service.
Evaluate the implementation by the proportion of families that initiate community services. | 12 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate whether families initiated participation in the community services to which they were referred, if any. This outcome will be measured as the proportion of families referred to community services that initiate participation in at lease one community service.
Evaluate the implementation by the proportion of families that initiate community services. | 24 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate whether families initiated participation in the community services to which they were referred, if any. This outcome will be measured as the proportion of families referred to community services that initiate participation in at lease one community service.
Evaluate the implementation by the proportion of families that initiate community services. | 36 months
  This will be collected from case report forms completed by the Navigators. On the CRFs, Navigators will indicate whether families initiated participation in the community services to which they were referred, if any. This outcome will be measured as the proportion of families referred to community services that initiate participation in at lease one community service.
Evaluate the implementation by the families' satisfaction with the Navigation program. | 3 months
  This will be measured via participant self-reports as the percentage of families that rate themselves as satisfied or very satisfied with their Navigation experience and the percentage of families that would recommend the program to other families.
Evaluate the implementation by the families' satisfaction with the Navigation program. | 15 months
  This will be measured via participant self-reports as the percentage of families that rate themselves as satisfied or very satisfied with their Navigation experience and the percentage of families that would recommend the program to other families.
Evaluate the implementation by the families' satisfaction with the Navigation program. | 27 months
  This will be measured via participant self-reports as the percentage of families that rate themselves as satisfied or very satisfied with their Navigation experience and the percentage of families that would recommend the program to other families.
Evaluate the implementation by the families' satisfaction with the Navigation program. | 39 months
  This will be measured via participant self-reports as the percentage of families that rate themselves as satisfied or very satisfied with their Navigation experience and the percentage of families that would recommend the program to other families.
Evaluate the impact of the Navigation program by reviewing child maltreatment. | 12 months
  This will be measured through Child Protective Services records via a comparison of the Navigation group and control group in their likelihood of having a substantiated or "services needed" case of maltreatment.
Evaluate the impact of the Navigation program by reviewing child maltreatment. | 24 months
  This will be measured through Child Protective Services records via a comparison of the Navigation group and control group in their likelihood of having a substantiated or "services needed" case of maltreatment.
Evaluate the impact of the Navigation program by reviewing child maltreatment. | 36 months
  This will be measured through Child Protective Services records via a comparison of the Navigation group and control group in their likelihood of having a substantiated or "services needed" case of maltreatment.
Evaluate the impact of the Navigation program by reviewing child maltreatment. | 48 months
  This will be measured through Child Protective Services records via a comparison of the Navigation group and control group in their likelihood of having a substantiated or "services needed" case of maltreatment.
Evaluate the impact of the Navigation program by reviewing child maltreatment. | 60 months
  This will be measured through Child Protective Services records via a comparison of the Navigation group and control group in their likelihood of having a substantiated or "services needed" case of maltreatment.
Evaluate the impact of the Navigation program by reviewing maternal health. | 3 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing maternal health. | 15 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing maternal health. | 27 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing maternal health. | 39 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing maternal health. | 51 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing maternal health. | 63 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores of their ratings of their overall health, depression symptoms, anxiety symptoms, and substance abuse symptoms.
Evaluate the impact of the Navigation program by reviewing child health and development. | 3 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing child health and development. | 15 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing child health and development. | 27 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing child health and development. | 39 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing child health and development. | 51 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing child health and development. | 63 months
  This will be measured from parent reports via a comparison of the Navigation and control groups' mean scores on ratings of their overall health, social-emotional development, and cognitive development.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 3 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 15 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 27 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 39 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 51 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing parent and parent-child relationships. | 63 months
  This will be measured from participant self-reports via a comparison of Navigation and control groups' mean scores on ratings of their knowledge of child development, parenting self-efficacy, parenting stress, parent discipline behavior, and parent attributions of child behavior.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 3 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 15 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 27 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 39 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 51 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.
Evaluate the impact of the Navigation program by reviewing family service receipt and children's connection to medical home. | 63 months
  Family services receipt will be measured from parent reports via a comparison of the Navigation and control groups' mean number of community services they have accessed since receiving Navigation/the control intervention. Connection to a medical home will be measured from parent report via a comparison of the Navigation and control groups' likelihood of having a primary care physician for their child.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dodge, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No